CLINICAL TRIAL: NCT05347472
Title: The Efficacy of Therapeutic Exercises Delivered by Smartphone Application for Urinary Incontinence Among Women: a Randomized Controlled Trial
Brief Title: The Efficacy of Therapeutic Exercises Delivered by Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Saddam Kanaan, Associate Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20210408
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): In this group, women will receive the smartphone application intervention that will include daily physical therapy exercises program
  Interventions: Other: Smartphone application
- Control group (Placebo Comparator): In this group, women will receive the sham application that includes information and general advice about UI only
  Interventions: Other: Sham Smartphone application

INTERVENTIONS:
Other: Smartphone application — the smartphone application intervention will consist daily physical therapy exercises program. The application will include all the videos about the exercises and all information about the repetition, frequency, intensity, and position.
  Arms: Experimental group
Other: Sham Smartphone application — ham application that includes information and general advice about UI only
  Arms: Control group

SUMMARY:
Therapeutic exercise has been shown to be effective in Urinary Incontinence management. However, there is a lack of physiotherapy services provided such necessary treatment. Moreover, mobile applications are becoming popular, and there are limited applications designed to help women with Urinary Incontinence. Consequently, no study investigated the effect of a smartphone application with specific exercises program for Urinary Incontinence management. Therefore, the aim of this study is to determine the effect of a Urinary Incontinence exercises delivered by smartphone application on UI outcomes.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a common health disorder among women in Jordan and worldwide. UI affects women's quality of life, mental health symptoms, and social participation. However, limited numbers of women with UI seek help for their problems for many reasons, including lack of rehabilitation services, feelings of shame, and unwillingness to discuss their problems. Therapeutic exercise has been shown to be effective in UI management. However, there is a lack of physiotherapy services provided such necessary treatment. Moreover, mobile applications are becoming popular, and there are limited applications designed to help women with UI. Consequently, no study investigated the effect of a smartphone application with specific exercises program for UI management. Therefore, the aim of the study is to develop an evidence-based therapeutic exercise application for UI and investigate its efficacy on UI clinical outcomes. We hypothesize that patients in the intervention group will have a significantly lower score of International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) , a lower score of perceived stress scale, lower Depression Anxiety and Stress scale (DASS-21) score, a higher score of Multidimensional Scale of Perceived Social Support (MSPSS), a higher Short Form Health Survey (SF-12) score, and a higher score of Incontinence Modular Questionnaire-Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) in comparison to the control group.

A randomized controlled trial design. Sixty women with urinary incontinence will be included in this study. Participants will be randomized to the intervention group who will receive the mobile application (will include general information about UI and exercises) and the intervention group who will receive the sham application (include information about UI only). Outcome measures will include Arabic ICIQ-UI SF to assess the frequency of urinary incontinence, the Arabic version of MSPSS to assess the social support, the Arabic version of (DASS-21) to assess the mental health symptoms, SF-12 to assess the quality of life, and ICIQ-LUTSqol to assess the quality of life of women with UI.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with UI, aged between 18-40, ability to read and own and use smartphone applications

Exclusion Criteria:

* Women with no medical diagnosis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with UI
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Modular Questionnaire-Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol). | Change from baseline to 4 weeks and 16 weeks
  The questionnaire assesses the quality of life of women with UI.
Arabic International Consultation on Incontinence Questionnaire-Urinary | Change from baseline to 4 weeks and 16 weeks
  Provides measurement of severity of UI and its impact on daily life
Arabic version of Multidimensional Scale of Perceived Social | Change from baseline to 4 weeks and 16 weeks
  Self-report measure of subjectively assessed social support

SECONDARY OUTCOMES:
Short Form Health Survey | Change from baseline to 4 weeks and 16 weeks
  Measures a person's health-related quality of life
Depression Anxiety Stress Scales | Change from baseline to 4 weeks and 16 weeks
  Measure the emotional state of depression, anxiety, and stress

CONTACTS AND LOCATIONS:
Overall Officials: Saddam F Kanaan, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: No